CLINICAL TRIAL: NCT05569200
Title: The Clinical Trial About Treatment of Benign Uterus Myoma by Haifu Focused Ultrasound Tumor Therapeutic System.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202111052RIPC
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Benign Uterine Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Haifu Focused Ultrasound tumor therapeutic System (Experimental)
  Interventions: Device: Haifu Focused Ultrasound tumor therapeutic System

INTERVENTIONS:
Device: Haifu Focused Ultrasound tumor therapeutic System — The device used in this trial will be Haifu Focused Ultrasound tumor therapeutic System. In Uterine benign tumor female, the investigators will observe the possibility of complication and tumor response of treatment.

SUMMARY:
Uterine benign tumor including myoma is the most common female benign pelvic tumor. Magnetic resonance-guided high-intensity focused ultrasound (MR-HIFU) has been considered to be a minimal invasive treatment. The device used in this trial will be Haifu Focused Ultrasound tumor therapeutic System. In this trial, the investigators will observe the possibility of complication and tumor response of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Benign uterine fibroids.
2. Women over the age of 20.
3. Abdominal circumference <100 cm.
4. The largest fibroids are ≥ 4 cm.

Exclusion Criteria:

1. Pregnant women or those with positive pregnancy test results.
2. Those with other pelvic diseases.
3. Those with immune diseases.
4. There are unsuitable interfaces in the ultrasonic treatment path.
5. Those with tumor calcification.
6. People with severe heart, blood vessel and kidney disease.
7. Those with abnormal coagulation function and low platelets.
8. Type III fibroids according to Funaki classification

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of tumour response | 3 month after treatment
  Evaluation of tumour response according to the modified RECIST criteria by sequencing MR imaging

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan